CLINICAL TRIAL: NCT00396552
Title: Treating Refractory Obsessive Compulsive Disorder With Repetitive Transcranial Magnetic Stimulation: A Double-blind Sham Controlled Longitudinal Study
Brief Title: Treating Refractory Obsessive Compulsive Disorder With rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Peggy Richter, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100/2006
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Obsessive Compulsive Disorder
Keywords: refractory transcranial magnetic stimulation; obsessive compulsive disorder; randomized; placebo-controlled; double-blind
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: refractory transcranial magnetic stimulation (rTMS)
- 2 (Sham Comparator)
  Interventions: Device: Sham condition

INTERVENTIONS:
Device: refractory transcranial magnetic stimulation (rTMS) — Bilateral rTMS will be delivered according to the following protocol: high frequency left (HFL) stimulation will initially be applied at 20 Hz, in 25 trains of 1.5 second duration with a 30 second interval between trains and at 100% of the RMT for a total of 25 minutes of stimulation. Following this HFR stimulation will be applied at the same parameters. Therefore a total of 50 minutes of stimulation will be delivered.
  Arms: 1
Device: Sham condition — Sham stimulation will be made at the site of active treatment but with only the side edge resting on the scalp. It will be administered as HFL and HFR for 50 minutes but with the coil angled 45-90 degrees away from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those with active stimulation but with minimal direct brain effects. Participants will be unable to see the stimulating coil and therefore will remain blind to the treatment condition.
  Arms: 2

SUMMARY:
Obsessive-compulsive disorder (OCD) is a severe psychiatric condition with only limited response to current first-line treatments, comprising pharmacotherapy and cognitive-behavioural therapy. Repetitive transcranial magnetic stimulation (rTMS) is a relatively new technique which has shown great promise in the treatment of refractory mood disorders, and schizophrenia, by alteration of brain activity. Previous work has demonstrated altered cortical excitability in OCD and preliminary studies have suggested that rTMS may have therapeutic potential in OCD. This pilot study will investigate the effectiveness of rTMS for treatment-refractory OCD, and establish appropriate treatment parameters. In addition, mechanisms whereby rTMS exerts its therapeutic effect will be explored using TMS to evaluate cortical inhibition and measures of cognitive biases and processing.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a severe and debilitating psychiatric illness characterized by intrusive unwanted thoughts (obsessions) and repetitive or ritualistic actions intended to reduce anxiety (compulsions). OCD is common with lifetime prevalence estimated at 2.5%, equally affecting both genders and all ethnic groups. It is also typically chronic in nature, resulting in substantial impact on quality of life. Functioning can be markedly impaired; it has been estimated that 20% of individuals with OCD should be considered severely affected. Although the pathophysiology is unclear, hyperactivity in the prefrontal orbital cortex has been consistently demonstrated, and normalizes with treatment. A decrease in cortical inhibition has been implicated in OCD utilizing a variety of methods, including paired-pulse TMS.

First-line treatment typically consists of either cognitive-behavioural therapy and/or pharmacotherapy with serotonin reuptake inhibitors (SSRI's or clomipramine). Ordinarily only modest benefits are obtained with conventional pharmacotherapy, with the majority of patients considered nonresponsive or only partially responsive. The limited success of conventional treatment makes identifying alternative treatments a priority. Although psychosurgery is regarded as a valid alternative for severe and refractory individuals, the potential for serious and irreversible adverse consequences is significant, rendering this a treatment of 'last resort' only. Repetitive TMS appears to represent a safe and effective alternative for severe sufferers.

Repetitive TMS has been shown to be an effective therapeutic tool for the treatment of several neuropsychiatric disorders including MDD and schizophrenia, but investigations into its utility in OCD are very preliminary. In a study of 12 OCD patients single session stimulation of the right lateral prefrontal cortex (20 Hz, 80% motor threshold, for 20 minutes) resulted in a decrease in compulsive urges for eight hours in contrast to the left prefrontal cortex which was associated with more modest response . Sachdev et al randomly assigned 12 individuals to receive right or left dorsolateral prefrontal stimulation (10 Hz,110% resting motor threshold, 15 minutes 5 sessions/week for 2 weeks). Subjects showed significant improvement at two weeks and 1-month follow-up, regardless of lateralit. A randomized controlled trial comparing right prefrontal stimulation to sham treatment in 18 OCD subjects was negative, however low frequency (1 Hz) stimulation was used in contrast to previous reports (110% motor threshold, 20 minutes 3 times/week for 6 weeks). Most recently a small study of 10 individuals with OCD and/or Tourette's syndrome found benefit with low-frequency stimulation of the supplementary motor area (1 Hz, 100% motor threshold, 20 minutes 5 sessions/week for 2 weeks). Notably subjects were treatment-resistant in both this and the Sachdev study. Thus although this limited literature precludes any definitive conclusions, it suggests that rTMS may be of benefit in refractory OCD.

In this study we propose to investigate the effectiveness of rTMS treatment in refractory OCD. Although ideal treatment parameters need to be established, the above literature suggests that high frequency stimulation of the dorsolateral prefrontal cortex is likely to be beneficial. Bilateral stimulation will be used; our previous work has demonstrated this method to be safe and well tolerated. Moreover patients will be assigned in randomized double-blind fashion to receive either active or sham TMS, allowing for more definitive conclusions to be drawn. We also propose to explore whether the induction of CI mediates the therapeutic effects of rTMS on OCD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* voluntary and competent to consent based on their ability to provide a spontaneous narrative description of the key elements of the study
* have a Structured Clinical Interview for DSM-IV (SCID) confirmed diagnosis of OCD
* are between the ages of 18 and 65
* have failed to achieve a clinical response, or did not tolerate, at least 3 separate antidepressant trials of sufficient dose for at least 10 weeks
* have a score of greater than or equal to 17 on the Y-BOCS. A careful medical and neurological history will be taken to ensure that subjects have no unstable conditions that would preclude them from entering into the study. This history will focus on conditions such as seizures, stroke, hypertension, diabetes, coronary artery disease, thyroid problems, respiratory illness, allergies and presence of metal implants

Exclusion Criteria:

* have a history of DSM-IV substance dependence in the last 6 months, and have DSM-IV substance abuse in the last month
* have a concomitant major unstable medical or neurologic illness or have had a history of seizures
* acutely suicidal
* are pregnant
* have metal implants. With respect to concomitant medications, patients will be excluded if they are currently (or in the last 4 weeks) taking: (a) more than lorazepam 2 mg daily (or equivalent), (b) monoamine oxidase inhibitors, (c) and/or bupropion due to its associated increased risk for seizures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Degree of change on the Yale-Brown Obsessive Compulsive Disorder Scale | intermittent

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Richter, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Background] Fitzgerald PB, Benitez J, de Castella A, Daskalakis ZJ, Brown TL, Kulkarni J. A randomized, controlled trial of sequential bilateral repetitive transcranial magnetic stimulation for treatment-resistant depression. Am J Psychiatry. 2006 Jan;163(1):88-94. doi: 10.1176/appi.ajp.163.1.88. PMID 16390894
- [Background] Loo CK, Mitchell PB. A review of the efficacy of transcranial magnetic stimulation (TMS) treatment for depression, and current and future strategies to optimize efficacy. J Affect Disord. 2005 Nov;88(3):255-67. doi: 10.1016/j.jad.2005.08.001. Epub 2005 Sep 2. PMID 16139895
- [Background] Klein E, Kolsky Y, Puyerovsky M, Koren D, Chistyakov A, Feinsod M. Right prefrontal slow repetitive transcranial magnetic stimulation in schizophrenia: a double-blind sham-controlled pilot study. Biol Psychiatry. 1999 Nov 15;46(10):1451-4. doi: 10.1016/s0006-3223(99)00182-1. PMID 10578460
- [Background] Hoffman RE, Hawkins KA, Gueorguieva R, Boutros NN, Rachid F, Carroll K, Krystal JH. Transcranial magnetic stimulation of left temporoparietal cortex and medication-resistant auditory hallucinations. Arch Gen Psychiatry. 2003 Jan;60(1):49-56. doi: 10.1001/archpsyc.60.1.49. PMID 12511172
- [Background] Greenberg BD, Ziemann U, Cora-Locatelli G, Harmon A, Murphy DL, Keel JC, Wassermann EM. Altered cortical excitability in obsessive-compulsive disorder. Neurology. 2000 Jan 11;54(1):142-7. doi: 10.1212/wnl.54.1.142. PMID 10636140
- [Background] Mantovani A, Lisanby SH, Pieraccini F, Ulivelli M, Castrogiovanni P, Rossi S. Repetitive transcranial magnetic stimulation (rTMS) in the treatment of obsessive-compulsive disorder (OCD) and Tourette's syndrome (TS). Int J Neuropsychopharmacol. 2006 Feb;9(1):95-100. doi: 10.1017/S1461145705005729. Epub 2005 Jun 28. PMID 15982444
- [Background] Sachdev PS, McBride R, Loo CK, Mitchell PB, Malhi GS, Croker VM. Right versus left prefrontal transcranial magnetic stimulation for obsessive-compulsive disorder: a preliminary investigation. J Clin Psychiatry. 2001 Dec;62(12):981-4. doi: 10.4088/jcp.v62n1211. PMID 11780880
- [Background] Horwath E, Weissman MM. The epidemiology and cross-national presentation of obsessive-compulsive disorder. Psychiatr Clin North Am. 2000 Sep;23(3):493-507. doi: 10.1016/s0193-953x(05)70176-3. PMID 10986723
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research